CLINICAL TRIAL: NCT05030454
Title: Pilot Study of a Novel Optical Surface Image Guidance System for Beam-Gated Online Adaptive SBRT Delivery in Mobile Lower Lung and Upper Abdominal Malignancies
Brief Title: Novel Optical Surface Image Guidance System for Beam-Gated Online Adaptive SBRT Delivery in Mobile Lower Lung and Upper Abdominal Malignancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202107198
Record Dates: First submitted 2021-08-19; First posted 2021-09-01 (Actual); Results first posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Any Solid Malignancies of Any Tissue Origin (Except for Small Cell Lung Cancer) Involving the Upper Abdomen and Thorax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- CT-guided stereotactic adaptive radiotherapy (Experimental): -Radiotherapy will consist of stereotactic body therapy, to be given over five fractions, delivered once daily or once every other day for a period of one to two weeks, for a total of five treatments.
  Interventions: Device: ETHOS; Radiation: CT-guided stereotactic adaptive radiotherapy

INTERVENTIONS:
Device: ETHOS — Ring-gantry CT-guided radiotherapy unit, pairing a linear accelerator within a ring-gantry imaging unit.
Radiation: CT-guided stereotactic adaptive radiotherapy — All participants will be initially planned to at least 35 Gy in 5 fractions, subject to hard constraints based on the treatment site.

SUMMARY:
Motion during radiation therapy can be categorized as inter-fraction (changes in anatomy that occur between treatment days) and intra-fraction (changes that occur during the "beam on" window of treatment delivery). Inter-fraction motion is managed by adaptive radiotherapy (ART), the process of making changes in the treatment plan while the patient remains on the treatment table. This is now a standard-of-care therapy within Washington University's clinic. Intra-fraction motion is managed by gated and non-gated delivery techniques. Varian Medical Systems has integrated the necessary components into a CT-guided radiotherapy device (ETHOS). In the ETHOS, Varian has built a device that integrates on-board cone beam CT imaging capable of delineating target and organ-at-risk positions and a dedicated artificial intelligence-driven treatment planning system for inter-fraction motion management as well as a paired optical surface image guidance system for intra-fraction motion management. Although online ART is a standard-of-care practice in the clinic and has previously been shown to be feasible, use of surface-guidance for intra-fraction gating of abdominal and thoracic SBRT on ETHOS is novel.

Therefore, in this study, the investigators propose to evaluate the feasibility and safety of using a novel surface guidance beam-gating system, incorporated with a CBCT-guided adaptive radiotherapy platform, to manage respiratory motion during delivery of CT-guided stereotactic radiotherapy. To best assess the utility of this technology to manage respiratory motion, the investigators will focus on disease sites that are highly affected by respiratory motion: upper abdominal or lower thoracic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Primary or metastatic disease of the abdomen or lower thorax, with biopsy-proven or radiographically diagnosed disease histology of solid tumor categorization, with the exception of small cell cancers.
* Must be medically fit for SBRT as determined by the treating physician, with at least one disease site to be deemed suitable for treatment with CT-guided stereotactic radiation to the abdomen or thorax as per radiation oncologist evaluation.
* At least 18 years of age.
* Karnofsky performance status > 60
* Capable of single deep inspiratory breath-hold or end-exhale breath-hold of at least 17 seconds in duration and of repeated end-exhale or deep inspiratory breath-hold of at least 10 seconds in duration upon verbal instruction.
* Must have completed any systemic therapy at least one week prior to planned start of SBRT (two weeks preferred), and must have no plans to initiate systemic therapy for at least one week following end of SBRT (two weeks preferred).
* Able to understand and willing to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Past history of radiotherapy within the projected treatment field of any of the disease sites to be treated by CT-guided SBRT.
* Currently receiving any investigational agents.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and/or breastfeeding. Patient must have a negative pregnancy test within 14 days of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Samson, M.D., MPHS, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) that will be used for individual participant data meta-analysis.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. Proposals may be submitted to the primary contact for this study.

REFERENCES:
- [Derived] Kiser K, Schiff J, Laugeman E, Kim T, Green O, Hatscher C, Kim H, Badiyan S, Spraker M, Samson P, Robinson C, Price A, Henke L. A feasibility trial of skin surface motion-gated stereotactic body radiotherapy for treatment of upper abdominal or lower thoracic targets using a novel O-ring gantry. Clin Transl Radiat Oncol. 2023 Oct 23;44:100692. doi: 10.1016/j.ctro.2023.100692. eCollection 2024 Jan. PMID 38021090
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CT-guided Stereotactic Adaptive Radiotherapy
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CT-guided Stereotactic Adaptive Radiotherapy
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 72 [40 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Scheduled Treatment Fractions Delivered Successfully Using the Surface Guidance System
Description: Success will be defined as delivery of a given treatment fraction in one on-table attempt, without requiring use of a secondary (backup) motion management system, or alternative treatment machine. Unsuccessful delivery of a fraction will be defined as multiple attempts for gating without reproducible positioning, breath-hold, and/or surface guidance feedback, such that the fraction is abandoned.
Time Frame: Through completion of treatment (estimated to be 2 weeks)
Measure: Number; unit: percentage of treatment fractions
Units Other Than Participants: Treatment fractions
Arm/Group | CT-guided Stereotactic Adaptive Radiotherapy
Number analyzed (Participants) | 10
Number analyzed (Treatment fractions) | 50
percentage of treatment fractions | 100

ADVERSE EVENTS:
Time Frame: Adverse events and all-cause mortality were tracked from start of treatment through 3 months following the last day of SBRT with the length of follow-up ranging from 3 months and 1 week for those who received their radiotherapy fraction daily or 3 months and 2 weeks for those who received their radiotherapy fraction every other day.
Arm/Group | CT-guided Stereotactic Adaptive Radiotherapy
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 2/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CT-guided Stereotactic Adaptive Radiotherapy (N=10)
Sepsis (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CT-guided Stereotactic Adaptive Radiotherapy (N=10)
Anorexia (Metabolism and nutrition disorders) | 1
Epigastric pain radiating to the back (Gastrointestinal disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Body aches (General disorders) | 1
Syncope (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-14): https://cdn.clinicaltrials.gov/large-docs/54/NCT05030454/Prot_SAP_000.pdf